CLINICAL TRIAL: NCT05851651
Title: The Effects and Experience of a Gestational Diabetes and Antenatal Human Milk Expression (GAME) Programme in Hong Kong Chinese Women
Brief Title: Gestational Diabetes and Antenatal Human Milk Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAME
Record Dates: First submitted 2023-04-17; First posted 2023-05-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-04

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care plus an antenatal milk expression education (Experimental): Participants will have one face-to-face breastfeeding education in lactation clinic at 37 weeks of gestation and telephone follow-up weekly till delivery.
  Interventions: Behavioral: Antenatal milk expression and breastfeeding self-efficacy enhancement
- Standard hospital antenatal care (No Intervention): Participants will receive standard care include prenatal breastfeeding education at gestation of 24-36 weeks same as intervention group. They will not discuss about antenatal milk expression, breastfeeding self-efficacy and the effects of breastfeeding on GDM women.

INTERVENTIONS:
Behavioral: Antenatal milk expression and breastfeeding self-efficacy enhancement — A face-to-face breastfeeding education in lactation clinic at 37 weeks of gestation will be arranged. The session will approximately last for 45minutes. GDM leaflet and GAME fact sheet are used to facilitate the teaching. The benefits of breastfeeding for women with GDM will be addressed. Maternal metabolic control, calories consumed, and weight loss are addressed for the extra benefits of breastfeeding for GDM women. The possible challenges of GDM on breastfeeding will be supported. The antenatal human milk expression will be taught by International Board-Certified Lactation Consultant. Participants will be encouraged to express colostrum twice daily for up to 10 minutes until admitted to hospital to give birth. They will receive a weekly phone follows up from 38 weeks before delivery and they can contact the researcher by phone in the information sheet if any questions.
  Arms: Standard care plus an antenatal milk expression education

SUMMARY:
Exclusive breastfeeding is global recognized as the optimal infant feeding. Hong Kong is committed to promoting, protecting and supporting the global movement for successful breastfeeding. Exclusive breastfeeding is especially strongly recommended and supported to the maternal history of Gestational Diabetes Mellitus (GDM). This study aims to examine the acceptability and feasibility of Antenatal human milk expression (AME) as breastfeeding intervention to improve breastfeeding for GDM women. The efficacy of AME practice on the breastfeeding exclusivity will also be investigated. It is hypothesized that AME will increase breastfeeding exclusivity compare with women receiving standard care, and will improve the breastfeeding self-efficacy and reduce depressive symptoms of women after birth.

DETAILED DESCRIPTION:
The incidence of GDM has been increasing worldwide and varied globally. Women with previous GDM have a 7-fold higher risk of developing diabetes mellitus over their lifetime. It has emerged global public health concern. Studies found that women with GDM breastfeed her baby significantly reduce the risk of Type 2 Diabetes and cardiometabolic disease, and improve postpartum glucose metabolism. However, evidence shows that GDM women have breastfeeding challenges and barriers. Women with diabetes experience delay in lactogenesis and infant have increased risk hypoglycaemia, they require blood monitoring and are often admit to the neonatal unit. As a result, the infants are more likely to have early receiving of formula supplementation. Besides, evidence indicated that low maternal confidence, increase depressive symptoms and breastfeeding self-efficacy among GDM women. Therefore, early lactation support was necessary. Greater support for GDM women reduces the risks of hypoglycaemia, formula supplementation and early weaning. It has been proposed that hand expression of breast milk in pregnancy may promote breastfeeding. Mothers with diabetes can express colostrum antenatally for use rather than infant formula if necessary.

Though Antenatal Milk Expression (AME) advises women at risk of early lactation problems, very limited evidence regarding the safety and efficacy of the practice. Also, very limited evidence investigated the AME for diabetes women for improving infant outcomes. Few studies found that AME increased confidence and contributed to better preparation on breastfeeding, but AME on depressive symptoms is under examined.

In Hong Kong, AME is not widely practice with inconsistent advice. It may raise concern on culture diversity regarding conservative culture in Chinese. There is lack of local article on the feasibility and acceptability of AME practice for GDM women in Hong Kong. Local clinical protocol on the implementation of AME and instructions on the practice is also absent. Given cultural differences in breastfeeding motivation and self-regulation as compared with those of oversea countries, the motivation of Hong Kong pregnant women engages in antenatal education and receiving social and breastfeeding support may be differ from women in the West. Thus, it is important to evaluate the efficacy and experience of AME on Hong Kong Chinese to assess cultural acceptability and effectiveness in supporting baby-friendly hospital practice and breastfeeding continuation.

Limited qualitative study compares breastfeeding self-efficacy on GDM women and positive impacts of the self-efficacy on breastfeeding prevalence and duration. Besides, qualitative study on the experiences and perceptions of GDM women on breastfeeding, and the experience on the collection and storage of expressed colostrum are very rare.

This blocked randomized, parallel-armed controlled trial with mixed method study design which integrating with quantitative and qualitative study will be conducted to examine (1) the acceptability and feasibility of AME as breastfeeding intervention to improve breastfeeding for GDM women, how and why AME works or does not work using qualitative research; (2) to understand the experience and perceptions of antenatal milk expression among the GDM women and (3) to investigate the efficacy of AME practice on the breastfeeding exclusivity. The secondary aims are determining whether AME as mediating variables in the effect on the breastfeeding self-efficacy among Hong Kong GDM women in Hong Kong.

The study hypotheses are (1) Antenatal human milk expression (AME) will increase breastfeeding exclusivity on hospital discharge, at 4 weeks and 8 weeks postpartum compare women receiving standard care (2) AME will improve the breastfeeding self-efficacy and reduce depressive symptoms of women after birth.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed gestational diabetes without on insulin
* can read and speak Chinese
* Hong Kong resident and stay in Hong Kong after delivery
* no serious medical or obstetrical complications
* no mental health illness or history
* have regular antenatal check-up
* singleton pregnancy
* primiparous or multiparous women
* intention to breastfeed
* pre-pregnancy BMI<25

Exclusion Criteria:

* do not have Hong Kong Identify Card
* breastfeeding elder child at pregnancy
* cannot understand the study
* give birth <37 weeks of gestation
* a known fetal anomaly or any suspicion of fetal compromise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Infant Feeding pattern | At 4 weeks postpartum
  Exclusive breastfeeding prevalence
Infant Feeding pattern | At 8 weeks postpartum
  Exclusive breastfeeding prevalence

SECONDARY OUTCOMES:
Women's self-determination toward breastfeeding | At baseline, 4 weeks and 8 weeks postpartum
  Chinese Breastfeeding Self -Regulation Questionnaire is a psychometric tested valid and reliable tool to measure maternal self-determination towards breastfeeding. The Cronbach's alpha of the BSRQ was 0.86. For every one-point increase in the BSRQ score, participants had 15% higher odds of any breastfeeding (OR=1.15, 95%CI 1.07-1.23) and 9% higher odds of exclusive breastfeeding (OR=1.09, 95%CI 1.02-1.17) at 6 weeks postpartum.
Women's self-efficacy in breastfeeding | At baseline, 4 weeks and 8 weeks postpartum
  Breastfeeding Self-Efficacy Scale-Short Form is used to measure maternal breastfeed confidence during postpartum. This instrument consists of 14 items, ranging from 1 = 'Not at all confident' to 5= 'Very confident.' The summary score from 14 to 70 is created by adding 14 items. The scale is psychometrically tested, demonstrates a consistent high reliability and validity. Low breastfeeding self- efficacy is significant predictor of early attrition of breastfeeding.
Women's perinatal/postnatal depression | At baseline, 4 weeks and 8 weeks postpartum
  Edinburgh Perinatal/Postnatal Depression Scale is used during antepartum and postpartum. It consist of 10 items include anxiety and depressive and symptoms; cut-off point is 9/10. It has a sensitivity of 0.86 and specificity of 0.78 with a positive predictive value of 73%. It psychometrically tested, high reliability and validity for perinatal and at 6 weeks postpartum. Successful breastfeeding is predictive of lower maternal depressive symptomology.
Women's prevalence of Impaired Glucose Tolerance | At 6 weeks postpartum
  Prevalence of IGT among participants according to breastfeeding status (any breastfeeding or exclusive formula feeding) will be collected from medical record for the fasting blood sugar testing at 6 weeks postpartum.

OTHER OUTCOMES:
Women's experience, perception, and attitude for AME practices | At 6 weeks postpartum
  Those participants response the highest and lowest self-efficacy score at baseline and 4 weeks postpartum will be invited to join the interview. The interview will last approximately 60-90 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Ngai Ms Leung, MPH, Principal Investigator — Department of Obstetrics and Gynaecology, Kwong Wah Hospital
Locations (2):
- Hong Kong (2):
  - Kwong Wah Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No